CLINICAL TRIAL: NCT00324688
Title: Open-label Multicenter Study to Assess the Efficacy, the Tolerability and the Adherence of a Once Daily (QD) Taken Antiretroviral Therapy (ART) Containing the NtRTI Tenofovir DF 300 mg in Combination With the Best Suitable Once a Day Regimen Being 1 NRTI Plus 1 PI or 1 NRTI Plus 1 NNRTI in HIV-1-infected IVDU- Patients With Opiate Substitution Being Either Antiretroviral-naive or With Suppressed Viral Load and Without a History of Virological Failure
Brief Title: Safety Study of Once a Day ART and Opiate Substitute.
Acronym: 3OD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-MC-104-1015; GS-02-1015
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Methadone; HIV-1 infection
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Viread

SUMMARY:
This study looks at HIV-infected subjects who are on methadone treatment and medicines for HIV.

DETAILED DESCRIPTION:
Patients with a history of opiate abuse (IVDU) are not only a patient population that is frequently difficult to reach by the healthcare system, but it also exhibits specific problems in HIV-treatment (ART). These patients frequently have a chaotic lifestyle, which makes it difficult to take medications regularly. Amongst the reasons for this are housing difficulties, intoxication and substance abuse.

The introduction of opiate substitution treatment can help to provide some structure and certainty to patients. Even so IVDU patients are often started on ART later than others and have a greater tendency to have treatment interruptions and sub-optimal adherence to ART. The end result can be treatment failure and the development of drug resistance.

There is an unmet medical need for ART regimens that make adherence easier and may be suitable for co-administration with once-daily opiate substitution.

The availability of tenofovir disoproxil fumarate (DF) 300 mg offers new options in the creation of once-daily regimens with reduced potential for drug-drug-interactions. It is believed that it is now possible to construct viable once daily HIV treatment regimens for patients who have either never received prior therapy or who have no history of drug resistance. Tenofovir DF is administered as a single 300 mg tablet once daily with food for the treatment of HIV infection. This once daily dosing schedule of tenofovir DF makes it an attractive option for simplified dosing regimens in many subjects, including methadone-maintained individuals infected with HIV. Because many opiate-maintained subjects are required to have their methadone dosing directly observed in the clinic, there is considerable interest in using directly-observed therapy (DOT) in such subjects. Given that tenofovir is eliminated renally and methadone is predominantly hepatically metabolized, the potential for a pharmacokinetic interaction is low. However, other antiretroviral agents with substantial renal elimination such as didanosine and stavudine have been shown to interact pharmacokinetically with methadone. Thus, it is important to demonstrate that tenofovir DF and methadone can be administered together safely and without concern for a pharmacokinetic interaction and/or alterations in the efficacy, safety, or tolerability of methadone maintenance such that dose modifications would be required. This can also be influenced by the other products in the combination therapy.

HIV/HBV coinfection is a frequent issue in this population (> 20%). Treatment with TDF, which is active against HBV, could help to stabilize the chronic HBV infection, even in cases with Lamivudine-resistance.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Previously documented diagnosis of HIV-1 infection:

  * by antibody assay (enzyme immunoassay confirmed by western immunoblot); or
  * positive HIV culture; or
  * detectable plasma HIV-1-RNA levels by reverse transcriptase polymerase chain reaction (RT-PCR).
* Receiving stable opiate substitution (stable methadone level for ≥ 2 weeks prior to entry into the study) with methadone, levomethadone or buprenorphine
* Either:

  * Antiretroviral (ARV) therapy-naïve(*) and with:

    * CD4 counts < 351 cells/µL; and/or
    * HIV-1 plasma levels >= 30,000 copies/mL (*)less than 3 months of ART for vertical transmission is considered as ARV therapy naïve.
  * Or restarting ART after treatment discontinuation with no evidence of prior HIV virological failure (virological failure defined as 2 consecutive measurements 4 weeks apart with viral load of HIV RNA > 400 copies/mL while on ART)
  * Or currently receiving stable ART therapy and with virological suppression (< 400 copies/mL), for at least 6 months and:

    * suffering from adherence problems because of dosing of current ART; or
    * suffering from side effects on the current recorded ART.
* Able to give informed consent
* In the opinion of the investigator is likely to be able to complete the study

Exclusion Criteria:

* Need for antiretroviral therapy which is not according to protocol
* Pregnant or breastfeeding women
* Females of childbearing potential not willing to use a barrier method(s) of contraception during heterosexual intercourse during the duration of the study
* Contraindication to use of tenofovir DF 300 mg or another concomitant medication
* Known hypersensitivity to the active component or excipients
* Prior receipt of tenofovir
* Evidence of clinical, genotypic, or phenotypic resistance to any ARV
* History of virological failure while on previously recorded ART regimens (virological failure defined as 2 consecutive measurements 4 weeks apart with viral load of HIV RNA > 400 copies/mL)
* Acute, life-threatening infection or malignancy that needs systemic therapy
* Any clinical laboratory findings obtained during screening that could be a risk factor for the patient during the study:

  * Grade 4 increase of any laboratory value
  * Grade 3 (> 5-10 upper limit of normal [ULN] increase in transaminases) at the screening visit
  * Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
* Current use of medication that, in the investigator's opinion or sponsor's opinion, will interfere with the study medication
* Participation in other clinical trials
* More than three months of ART treatment for vertical transmission prophylaxis
* Current receipt of adefovir dipivoxil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-03; Study Completion 2006-06

PRIMARY OUTCOMES:
Proportion of patients with HIV RNA < 400 and with HIV RNA < 50 copies/mL at Week 48

SECONDARY OUTCOMES:
Proportion of patients with HIV RNA < 400 and with HIV RNA < 50 copies/mL at Week 24
Time to failure or ART discontinuation. Virological failure is defined as 2 consecutive measurements 4 weeks apart with viral load of HIV RNA > 400 copies/mL
Adherence to HIV treatments (Medication Adherence Self-Report Inventory [MASRI] questionnaire, monthly evaluation through patient diary)
Adherence to opiate substitution treatment
Correlation of adherence to ART and HIV RNA levels
Percentage of patients with HIV-1 RNA below limit of detection < 400 copies/mL and 50 copies/mL and adherence level > 95%, > 90%, > 85%, > 80%, > 75%, > 70%, > 50% and < 50%
Dose adjustments for methadone
Proportion of patients with any adverse event (AE)/serious adverse event (SAE)
Proportion of patients with AE/SAE classified by body system
Proportion of patients with each AE/SAE
Distribution of intensity of each AE/SAE (the highest intensity per patient for each event will be considered)
Distribution of relationship to study drug (the strongest relationship to study drug per patient for each event will be considered)
Distribution of toxicity grade (the highest grade per patient for each test will be considered)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mertenskoetter, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Munich, Germany